CLINICAL TRIAL: NCT04561232
Title: Locomotor Learning in Infants at High Risk for Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Hospital Los Angeles (Other); University of Oklahoma (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-016773; 1R01HD098364-01A1 (NIH)
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; infant; physical therapy; motor learning; robotics
MeSH Terms: conditions — Cerebral Palsy | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Locomotor Learning (Other): This study has three phases. The first phase of the study will be the observation of early spontaneous leg movements which will be measured monthly from 1-4 months of age.
  The prone locomotor intervention phase using the Self-Initiated Prone Progression Crawler (SIPPC) will occur from 5-9 months of post-term age, or end earlier if the child achieves the ability to crawl six feet. Treatment will occur at an intensity of 3 times per week for 15-30 minutes. Infants will use the SIPPC for the duration of each therapy session
  The upright locomotor intervention phase using DWS will occur from 9-18 months of age, or begin earlier if the child achieves the ability to crawl six feet before 9 months of age, and end earlier if the child achieves independent walking before 18 months of age. Treatment will occur at an intensity of 3 times per week for 30 minutes. Infants will receive dynamic weight support (DWS) for the duration of the 30-minute therapy session.
  Interventions: Behavioral: Prone and Upright Locomotor Training

INTERVENTIONS:
Behavioral: Prone and Upright Locomotor Training — During the movement observation phase, infants will wear a wireless movement sensor at each ankle for two days. Research staff will show the caregivers how to place the sensors in the morning and charge them overnight.
  The training protocol for the prone training will consist of: 1) Warm-up. 2) Assisted movement of the arms and legs. 3) Calibration of the infant's arm and leg positions. 4) Self-initiated mobility for up to five minutes.
  For upright training, the environment will be arranged to encourage active motor exploration and variability in walking activities.The therapist will assist the child as needed to encourage upright locomotor activities, but only the minimum amount needed to perform the task. Weight assistance will be gradually reduced as postural control and coordination improve.
  Other Names: Crawling therapy; Walking therapy

SUMMARY:
The objective of this project is to characterize the evolution of locomotor learning over the first 18 months of life in infants at high risk for cerebral palsy (CP). To characterize how locomotor skill is learned (or not learned) during this critical period, the investigators will combine established protocols using robust, unbiased robotic and sensor technology to longitudinally study infant movement across three consecutive stages during the development of impaired human motor control - early spontaneous movement, prone locomotion (crawling), and upright locomotion (walking).

DETAILED DESCRIPTION:
Early spontaneous leg movements will be measured monthly from 1-4 months of age. Infants who remain at high risk for CP by month 4 as measured by the General Movements Assessment and the Test of Infant Motor Performance (TIMP) at 4 months of age will continue to locomotor training phases. Prone locomotor training using the Self-Initiated Prone Progression Crawler (SIPPC) will be delivered from 5-9 months of age. Upright locomotor training with dynamic weight support (DWS) will be delivered from 9-18 months of age. Repeated assessments of locomotor skill, movement quality, training characteristics, and variables that may mediate locomotor learning will be collected at time points from 1 month to 18 months of post-term age.

Investigators will examine the relationships between motor error and locomotor skill acquisition over time, anticipating that experiencing and correcting movement errors is critical to skill acquisition in infants at risk for CP; the contribution of other training characteristics (movement time, movement variability, and postural control) to locomotor learning; and how learning is mediated by neurobehavioral factors outside of training. Investigators will develop comprehensive models of training predictors and mediators for prone and upright locomotor learning.

ELIGIBILITY:
Inclusion Criteria:

* less than 6 weeks of age (corrected for prematurity, if applicable)
* have a history of an early brain injury associated with high risk for cerebral palsy including periventricular leukomalacia, hypoxic-ischemic encephalopathy, intraventricular hemorrhage, hydrocephalus, stroke, neonatal seizures, or intracranial cystic lesion
* family is able to commit to study visits

Exclusion Criteria:

* known genetic condition unrelated to cerebral palsy (CP) or congenital abnormalities

Infants with fidgety movements on the General Movements Assessments (GMA) at 3 months of age or a score greater than -0.5sd below the mean on the Test of Infant Motor Performance at 4 months of age will not progress in the study because these infants are unlikely to have CP.

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-66 | Up to 18 months
  The Gross Motor Function Measure-66 (GMFM-66) is a Rasch-analyzed measure of gross motor function designed for children with cerebral palsy (CP). Computation of the GMFM-66 score involves statistical weighting of the raw item scores for difficulty. Scores range from 0 to 100 with higher scores indicating more functional ability.
Movement Observation Coding System | Up to 18 months
  The Movement Observation Coding System will use video coding to assess postural control, arm and leg movements, and goal directed movement.

SECONDARY OUTCOMES:
Early spontaneous movement | Up to 4 months
  Wearable sensor data will be analyzed to describe leg movements produced across in the natural environment.
Error rate - prone | Up to 18 months
  Error during prone locomotor training will measured using the Self-Initiated Prone Progression Crawler (SIPPC).
Error rate - upright | Up to 18 months
  Error during upright locomotor training will measured using the dynamic weight support (DWS) technology.
Movement index | Up to 18 months
  Movement index is the percent of time moving during each therapy session which will be recorded by sensors.
Postural control | Up to 18 months
  Postural control will be measured from video coding of therapy sessions.
Movement variability - prone | Up to 18 months
  Movement variability during prone locomotor training will be measured using the Self-Initiated Prone Progression Crawler (SIPPC).
Movement variability - upright | Up to 18 months
  Movement variability during upright locomotor training will be measured by video coding.

OTHER OUTCOMES:
Cognition | Up to 18 months
  The cognition age equivalent obtained from the Bayley Scales of Infant and Toddler Development- Fourth Edition (BSID-IV). This value describes what age the child is currently similar to in their cognitive performance, and all values are reported in months of age. The range of values on the scale 0-42 months of age. A higher number value means a greater cognitive ability.
Motivation to Move Scale | Up to 18 months
  The Motivation to Move Scale is scored from video data of infant behavior during treatment sessions. Children are classified on a scale of 1 to 5 with higher scoring indicating increased motivation to move.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Prosser, PhD, Principal Investigator — Research Scientist
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Pierce SR, Skorup J, Kolobe THA, Smith BA, Prosser LA. Agreement Between the Gross Motor Ability Estimator-2 and the Gross Motor Ability Estimator-3 in Young Children With Cerebral Palsy. Pediatr Phys Ther. 2024 Jan 1;36(1):37-40. doi: 10.1097/PEP.0000000000001065. Epub 2023 Nov 30. PMID 38033276
- [Derived] Prosser LA, Skorup J, Pierce SR, Jawad AF, Fagg AH, Kolobe THA, Smith BA. Locomotor learning in infants at high risk for cerebral palsy: A study protocol. Front Pediatr. 2023 Feb 23;11:891633. doi: 10.3389/fped.2023.891633. eCollection 2023. PMID 36911033

DOCUMENTS (1):
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT04561232/ICF_000.pdf